CLINICAL TRIAL: NCT05332340
Title: Phase 1 Clinical Trial Study to Evaluate Pharmacokinetics and Safety Profile of BZ371A in a Gel Formulation, Applied on Healthy Men and Women Genitals
Brief Title: Safety, Tolerability and Pharmacokinetics (PK) Evaluation of BZ371A, Topically Administered
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biozeus Biopharmaceutical S.A. (Industry)
Collaborators: Azidus Brasil Scientific Research and Development Ltda (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BZ371CLI003
Record Dates: First submitted 2022-02-22; First posted 2022-04-18 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Erectile Dysfunction Following Radical Prostatectomy; Erectile Dysfunction; Prostate Cancer; Radical Prostatectomy
Keywords: Erectile Dysfunction; Radical Prostatectomy; Prostate Cancer
MeSH Terms: conditions — Erectile Dysfunction; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Patients (Experimental): Healthy patients receiving topical application of BZ371A
  Interventions: Drug: BZ371A

INTERVENTIONS:
Drug: BZ371A — Single dose topical administration of 1.5 mL with a concentration of 5 mg/mL of BZ371A.

SUMMARY:
The purpose of this study is to evaluate pharmacokinetics, safety and tolerability profile of BZ371A topically administered in healthy patients.

DETAILED DESCRIPTION:
Prostate cancer remains one of the most prevalent cancer in men. For its treatment, recent technological advances demonstrate that the most effective treatment is the Radical Prostatectomy (RP) procedure. However, although curative for Prostate Cancer, can result in damage to the cavernosal nerves.

The cavernosal autonomic nerves travel posterolaterally to the prostate to enter the penis and regulate blood flow and hence erection. Thus, damage caused by RP will affect NO tissue release and blood flow regulation, causing erectile dysfunction.

BZ371A has the ability to restore local blood flow regulation by a new and innovative mechanism of action and, therefore, has potential to be a supportive therapy for RP patients (restoring the erectile function).

Thus, this study has the purpose to evaluate safety, tolerability and pharmacokinetics of a BZ371A single dose, topically administrated at the genital area.

ELIGIBILITY:
Inclusion Criteria:

* Men or women
* Body mass index > 19 and < 28.5 Kg/m2
* Is able to understand the Informed Consent Form (ICF)

Exclusion Criteria:

* Women in their menstrual period;
* Diseases that interfere with the absorption, distribution and excretion of drugs, such as history or presence of hepatic or renal diseases;
* Presence of active genital lesions or sexually transmitted disease (STD) (such as herpes, gonorrhea, candidiasis, Human Papillomavirus, and others) that impair analysis of local adverse effects on the genitalia;
* History of symptomatic hypotension, or diseases that increase the risk of symptomatic hypotension, such as patients with heart disease (including a history of angina and/or heart failure) and nephropathies;
* Findings on ECG and/or laboratory tests that, in the investigator's judgment, are considered the research volunteer's participation or may interfere with the analysis of the study of the study;
* Blood pressure (BP) outside the limits considered safe: systolic BP (SBP) 90 - 140 mmHg and diastolic BP diastolic BP (DBP) 60 - 90 mmHg, except for situations such as "white coat syndrome";
* Any disease or condition or physical finding that the investigator considers significant and that increases the risk
* Any disease or condition or physical finding that the investigator considers significant and that increases the risk of participation of the research volunteer or may interfere with the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Regina M Doi, Principal Investigator — Azidus Brasil Pesquisa Científica e LTDA
Locations (1):
- Azidus Brasil Pesquisa Científica e Desenvolvimento, Valinhos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Patients
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Patients
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years]
  Healhty Participants | 39.30 (9.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 3
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: Peak Plasma Concentration
Time Frame: 0 (Pre-dose), 15, 30, 60, 180 and 360 minutes post dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Healthy Patients
Number analyzed (Participants) | 12
ng/mL | NA (NA) — Below the level of detection

2. Primary Outcome: T1/2
Description: Terminal half-life of BZ371A
Time Frame: 0 (Pre-dose), 15, 30, 60, 180 and 360 minutes post dose
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Healthy Patients
Number analyzed (Participants) | 12
minutes | NA (NA) — Below the level of detection

3. Primary Outcome: AUC
Description: Area under the curve (AUC) of plasma/serum/blood drug concentration-time curve
Time Frame: 0 (Pre-dose), 15, 30, 60, 180 and 360 minutes post dose
Measure: Mean (Standard Deviation); unit: ng*min
Arm/Group | Healthy Patients
Number analyzed (Participants) | 12
ng*min | NA (NA) — Below the level of detection

4. Primary Outcome: Clearance (CL)
Description: Clearance of BZ371A
Time Frame: 0 (Pre-dose), 15, 30, 60, 180 and 360 minutes post dose
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Healthy Patients
Number analyzed (Participants) | 12
mL/min | NA (NA) — Below the level of detection

5. Primary Outcome: Vd
Description: Distribution Volume of BZ371A
Time Frame: 0 (Pre-dose), 15, 30, 60, 180 and 360 minutes post dose
Measure: Mean (Standard Error); unit: mL
Arm/Group | Healthy Patients
Number analyzed (Participants) | 12
mL | NA (NA) — Below the level of detection

6. Primary Outcome: Adverse Effects Evaluation
Description: Number of Adverse Effects after compound application
Time Frame: All adverse effect will be collected from the beginning of the study up to one week after drug administration
Measure: Number; unit: adverse events
Arm/Group | Healthy Patients
Number analyzed (Participants) | 12
adverse events | 2

7. Primary Outcome: Physical Exam
Description: Number of participants with abnormal physical exam findings
Time Frame: Baseline and 1 week
Measure: Number; unit: participants
Arm/Group | Healthy Patients
Number analyzed (Participants) | 12
participants | 0

8. Primary Outcome: Change in SBP
Description: Number of participants with a significant change in Systolic Blood Pressure
Time Frame: Baseline and 1 week
Measure: Number; unit: participants
Arm/Group | Healthy Patients
Number analyzed (Participants) | 12
participants | 1

9. Primary Outcome: Change in DBP
Description: Number of participants with a significant change in Diastolic Blood Pressure
Time Frame: Baseline and 1 week
Measure: Number; unit: participants
Arm/Group | Healthy Patients
Number analyzed (Participants) | 12
participants | 2

10. Primary Outcome: Change in Heart Rate
Description: Change in Heart Rate (HR).
  The data from this measure reflect changes calculated from the baseline.
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Healthy Patients
Number analyzed (Participants) | 12
bpm | 69.42 (12)

11. Primary Outcome: Change in Respiratory Rate
Description: Change in Respiratory Rate (RR).
  The data from this measure reflect changes calculated from the baseline.
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Healthy Patients
Number analyzed (Participants) | 12
breaths per minute | 19 (1)

12. Primary Outcome: Change in Temperature
Description: Temperature measurements.
  The data from this measure reflect changes calculated from the baseline.
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Healthy Patients
Number analyzed (Participants) | 12
degrees Celsius | 0.1 (0.36)
Statistical Analysis 1: Comparison: Healthy Patients; Test type: Superiority; p = 0.683, Kruskal-Wallis; Mean Difference (Final Values) = 0.1

13. Primary Outcome: Basal Chest Electrocardiogram (ECG)
Description: Number of participants with abnormal ECG readings
Time Frame: Baseline and 1 week
Measure: Number; unit: participants
Arm/Group | Healthy Patients
Number analyzed (Participants) | 12
participants | 0

14. Primary Outcome: Blood Evaluation
Description: Number of participants with abnormal laboratory test results
Time Frame: Baseline and 1 day
Measure: Number; unit: participants
Arm/Group | Healthy Patients
Number analyzed (Participants) | 12
participants | 0

15. Primary Outcome: Urine Evaluation
Description: Number of participants with abnormal urinalysis
Time Frame: Baseline and 1 week
Measure: Number; unit: participants
Arm/Group | Healthy Patients
Number analyzed (Participants) | 12
participants | 0

ADVERSE EVENTS:
Time Frame: 0 to 7 days from compound application
Description: 2 participants demonstrated mild Hypotension and 1 participant demonstrated Herpes labialis
Arm/Group | Healthy Patients
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Patients (N=12)
Hypotension (Vascular disorders) | 2 (2) — Non-symptomatic hypotension, with complete and spontaneous resolution
Herpes Labialis (General disorders) | 1 (1) — Herpes labialis was of moderate intensity

LIMITATIONS AND CAVEATS:
There were no relevant limitations and caveats to study execution

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/40/NCT05332340/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/40/NCT05332340/ICF_001.pdf